CLINICAL TRIAL: NCT00833027
Title: A 24 Week, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Adding Sitagliptin 100 mg Once Daily in Patients With T2DM Who Have Inadequate Glycemic Control on Metformin Therapy
Brief Title: ALPHA Sitagliptin Add on to Metformin (0431-103)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0431-103; MK0431-103; 2009_527
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Sitagliptin
  Interventions: Drug: sitagliptin phosphate

INTERVENTIONS:
Drug: sitagliptin phosphate — Sitagliptin 100 mg/day - tablet for 24 weeks
  Other Names: Januvia

SUMMARY:
Canadian physicians to experience in real life clinical practice the efficacy and tolerability of adding sitagliptin to their patients who have their glycemic levels inadequately controlled while on metformin

ELIGIBILITY:
Inclusion Criteria:

Patient Is Currently On Monotherapy With Metformin For At Least 10 Weeks Prior To Study Entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2009-10-30 (Actual); Study Completion 2009-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: 11-MAR-2008
  Last patient out: 30-OCT-2009
  Total number of sites: 110
Period: Overall Study
Arm/Group | Sitagliptin 100mg
Started | 608
Completed | 397
Not Completed | 211
Not completed — Adverse Event | 33
Not completed — Death | 1
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 24
Not completed — Protocol Violation | 115
Not completed — Withdrawal by Subject | 16
Not completed — Missing | 10

BASELINE CHARACTERISTICS:
Arm/Group | Sitagliptin 100mg
Number analyzed (Participants) | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258
  Male | 350
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 491
  Black | 16
  Hispanic | 6
  Asian | 73
  Native Indian | 6
  Other | 16
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent] | 7.73 (1.11)
Weight [Mean (Standard Deviation); unit: Kilograms] | 92.6 (24.42)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 9.3 (2.87)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24
Description: HbA1c is measured as percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent
Time Frame: Baseline and Week 24
Population: Includes all patients who received at least one dose of study medication and have a Week 24 measure.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sitagliptin 100mg
Number analyzed (Participants) | 375
Percent | -0.6 (0.95)
Statistical Analysis 1: Comparison: Sitagliptin 100mg; Test type: Superiority or Other; p < 0.001, Student's T-test; Student's T-test for paired samples; Mean Difference (Net) = -0.6, Standard Deviation 0.85

2. Secondary Outcome: Change From Baseline in HbA1c at Week 12
Description: HbA1c is measured as percent. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the Week 0 HbA1c percent
Time Frame: Baseline and Week 12
Population: Includes all patients who received at least one dose of study medication and have a Week 12 measure.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Sitagliptin 100mg
Number analyzed (Participants) | 406
Percent | -0.6 (0.85)

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100mg
Serious Adverse Events (participants affected / at risk) | 17/608
Other Adverse Events (participants affected / at risk) | 0/608
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100mg (N=608)
Acute coronary syndrome (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Sudden death (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.